CLINICAL TRIAL: NCT00735267
Title: A 52-Week Open-Label Safety Study of PD 0332334 in Subjects With Generalized Anxiety Disorder
Brief Title: A 52-Week Open-Label Safety Study of PD 0332334 in Subjects With Generalized Anxiety Disorder (GAD)
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Please see Detailed Description for termination reason.
Sponsor: Pfizer (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer, Inc.
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: A5361022
Record Dates: First submitted 2008-08-12; First posted 2008-08-14 (Estimated); Last update posted 2012-11-16 (Estimated); Status verified 2012-11

CONDITIONS: Generalized Anxiety Disorder
Keywords: Generalized Anxiety Disorder
MeSH Terms: conditions — Generalized Anxiety Disorder | interventions — imagabalin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: PD 0332334 — Dosage Form: 25 or 100 mg oral capsules Dosage and frequency: 350-600 mg twice a day Duration: 1 year
  Other Names: imagabalin

SUMMARY:
This study will assess the long-term safety and tolerability of 350 to 600 mg/day of PD 0332334 administered in split dose (twice daily) in subjects with Generalized Anxiety Disorder.

DETAILED DESCRIPTION:
Termination reason: On February 23rd 2009, a decision to terminate further development for PD 0332334 was communicated to investigators in this study. The decision to terminate this study was not based on any safety concerns.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must have completed all phases of one of the four preceding double-blind GAD studies.
* Female must continue to use adequate birth control methods and have a negative serum pregnancy test within 14 days prior to starting open label treatment.

Exclusion Criteria:

* Subjects who experienced a serious adverse event during the preceding double-blind efficacy study that was judged to be related to study medication by the investigator or the sponsor's medical monitor.
* Individuals who have an ongoing, unresolved, clinically significant medical problem that, in the judgment of the investigator or the sponsor's medical monitor, would make it unsafe for the subject to participate in the study.
* Serious suicidal risk per the clinical investigators's judgement.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 468 (Actual)
Dates: Start 2008-10; Primary Completion 2009-04 (Actual); Study Completion 2009-04 (Actual)

PRIMARY OUTCOMES:
The nature, incidence, and duration of adverse events monitored throughout the study by physical exam | Screening, Wk 25 & Wk 52/EOT
Electrocardiogram will be performed at screening and during follow up visits to assess the safety and tolerability of the compound in terms of clinically significant cardiovascular changes | Screening, Wk 4, Wk 25, Wk 52/EOT
The Columbia Suicide Severity Rating scale will be used to assess any suicide related adverse events | As needed
The nature, incidence, and duration of adverse events monitored throughout the study by vital signs evaluation at each visit, weight measurements and clinical laboratory monitoring periodically | Screening, Baseline, Wk 4, Wk 12, Wk 25, Wk 38, & Wk 52/EOT
All discontinuations due to adverse events will be reviewed throughout the trial to assess the safety and tolerability of the compound | Weekly

SECONDARY OUTCOMES:
The Hamilton Rating Scale for Anxiety (HAM-A) will be used to assess symptoms of Generalized Anxiety Disorder (GAD) over a one year time period. | Baseline, Wk 12, Wk 25, Wk 38, Wk 51 & Wk 52/EOT
The Clinical Global Impression of Severity (CGI-S), and the Daily Diary (DD) will also be used to assess symptoms of GAD over a one year time period. | Baseline, Wk 51 & Wk 52/EOT
The Health Care Utilization Questionnaire will be utilized to assess overall Health Care over a one year time period. | Baseline, Wk 12, Wk 25, Wk 38 & Wk 51

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (82):
- United States (82):
  - Pfizer Investigational Site, Birmingham, Alabama
  - Pfizer Investigational Site, Litchfield Park, Arizona
  - Pfizer Investigational Site, Arcadia, California
  - Pfizer Investigational Site, Beverly Hills, California
  - Pfizer Investigational Site, Costa Mesa, California
  - Pfizer Investigational Site, Encino, California
  - Pfizer Investigational Site, Escondido, California
  - Pfizer Investigational Site, Murrieta, California
  - Pfizer Investigational Site, National City, California
  - Pfizer Investigational Site, Newport Beach, California
  - Pfizer Investigational Site, Orange, California
  - Pfizer Investigational Site, Pasadena, California
  - Pfizer Investigational Site, Redlands, California
  - Pfizer Investigational Site, San Diego, California
  - Pfizer Investigational Site, Sherman Oaks, California
  - Pfizer Investigational Site, Temecula, California
  - Pfizer Investigational Site, Upland, California
  - Pfizer Investigational Site, Wildomar, California
  - Pfizer Investigational Site, Denver, Colorado
  - Pfizer Investigational Site, Hamden, Connecticut
  - Pfizer Investigational Site, Norwich, Connecticut
  - Pfizer Investigational Site, Altamonte Springs, Florida
  - Pfizer Investigational Site, Fort Myers, Florida
  - Pfizer Investigational Site, Jacksonville, Florida
  - Pfizer Investigational Site, Maitland, Florida
  - Pfizer Investigational Site, Miami, Florida
  - Pfizer Investigational Site, Orange City, Florida
  - Pfizer Investigational Site, Orlando, Florida
  - Pfizer Investigational Site, South Miami, Florida
  - Pfizer Investigational Site, West Palm Beach, Florida
  - Pfizer Investigational Site, Atlanta, Georgia
  - Pfizer Investigational Site, Marietta, Georgia
  - Pfizer Investigational Site, Libertyville, Illinois
  - Pfizer Investigational Site, Naperville, Illinois
  - Pfizer Investigational Site, Park Ridge, Illinois
  - Pfizer Investigational Site, Greenwood, Indiana
  - Pfizer Investigational Site, Terre Haute, Indiana
  - Pfizer Investigational Site, Overland Park, Kansas
  - Pfizer Investigational Site, Prairie Village, Kansas
  - Pfizer Investigational Site, Wichita, Kansas
  - Pfizer Investigational Site, Owensboro, Kentucky
  - Pfizer Investigational Site, Lake Charles, Louisiana
  - Pfizer Investigational Site, Baltimore, Maryland
  - Pfizer Investigational Site, Belmont, Massachusetts
  - Pfizer Investigational Site, Boston, Massachusetts
  - Pfizer Investigational Site, Fall River, Massachusetts
  - Pfizer Investigational Site, Haverhill, Massachusetts
  - Pfizer Investigational Site, Pittsfield, Massachusetts
  - Pfizer Investigational Site, Omaha, Nebraska
  - Pfizer Investigational Site, Las Vegas, Nevada
  - Pfizer Investigational Site, Nashua, New Hampshire
  - Pfizer Investigational Site, Albuquerque, New Mexico
  - Pfizer Investigational Site, Brooklyn, New York
  - Pfizer Investigational Site, New York, New York
  - Pfizer Investigational Site, Rochester, New York
  - Pfizer Investigational Site, The Bronx, New York
  - Pfizer Investigational Site, Raleigh, North Carolina
  - Pfizer Investigational Site, Columbus, Ohio
  - Pfizer Investigational Site, Dayton, Ohio
  - Pfizer Investigational Site, Toledo, Ohio
  - Pfizer Investigational Site, Bethany, Oklahoma
  - Pfizer Investigational Site, Oklahoma City, Oklahoma
  - Pfizer Investigational Site, Portland, Oregon
  - Pfizer Investigational Site, Salem, Oregon
  - Pfizer Investigational Site, Allentown, Pennsylvania
  - Pfizer Investigational Site, Media, Pennsylvania
  - Pfizer Investigational Site, Norristown, Pennsylvania
  - Pfizer Investigational Site, Philadelphia, Pennsylvania
  - Pfizer Investigational Site, Lincoln, Rhode Island
  - Pfizer Investigational Site, Columbia, South Carolina
  - Pfizer Investigational Site, Memphis, Tennessee
  - Pfizer Investigational Site, Austin, Texas
  - Pfizer Investigational Site, Dallas, Texas
  - Pfizer Investigational Site, DeSoto, Texas
  - Pfizer Investigational Site, Houston, Texas
  - Pfizer Investigational Site, Lake Jackson, Texas
  - Pfizer Investigational Site, San Antonio, Texas
  - Pfizer Investigational Site, Woodstock, Vermont
  - Pfizer Investigational Site, Charlottesville, Virginia
  - Pfizer Investigational Site, Seattle, Washington
  - Pfizer Investigational Site, Middleton, Wisconsin
  - Pfizer Investigational Site, Waukesha, Wisconsin

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A5361022&StudyName=A%2052-Week%20Open-Label%20Safety%20Study%20of%20PD%200332334%20in%20Subjects%20with%20Generalized%20Anxiety%20Disorder%20%28GAD%29